CLINICAL TRIAL: NCT06962774
Title: A Phase 1, Open-label, Single-dose Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics of a Single Oral Dose of ESK-001
Brief Title: An Investigational Study of ESK-001 in Participants With Normal Renal Function and Participants With Mild, Moderate, and Severe Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alumis Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESK-001-023
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healthy Volunteer (Experimental): Up to 24 healthy volunteer participants will receive a single dose of ESK-001
  Interventions: Drug: ESK-001
- Mild Renal Impairment (Experimental): 8 participants with mild renal impairment will receive a single dose of ESK-001
  Interventions: Drug: ESK-001
- Moderate Renal Impairment (Experimental): 8 participants with moderate renal impairment will receive a single dose of ESK-001
  Interventions: Drug: ESK-001
- Severe Renal Impairment (Experimental): 8 participants with severe Renal impairment will receive a single dose of ESK-001
  Interventions: Drug: ESK-001

INTERVENTIONS:
Drug: ESK-001 — Single oral dose of ESK-001 in participants from all cohorts

SUMMARY:
This a phase 1, open label, single dose, parallel cohort study to determine the pharmacokinetics (PK) of study drug (ESK-001) in healthy volunteer participants, and participants with mild, moderate, and severe renal impairment.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4) (A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.)

ELIGIBILITY:
Key Inclusion Criteria for All Participants:

* Body mass index between 18.0 and 40.0 kg/m2

Key Inclusion Criteria for Participants with Renal Impairment:

* Diagnosis of chronic, stable renal function in the 6 months prior to dosing, as determined by the investigator, based on medical history or eGFR, and not requiring dialysis

Key Exclusion Criteria for All Participants:

* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy, cholecystectomy, and hernia repair are allowed).

Key Exclusion Criteria for Participants with normal Renal function:

-Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator or designee.

Key Exclusion Criteria for Participants with Renal Impairment:

- History of any uncontrolled or unstable hepatic, hematological, gastrointestinal, neurological, endocrine, or psychiatric disorder, as determined by the investigator or designee, within 6 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | 48 hours
Incidence of nonserious adverse events (AE), serious adverse events (SAE), and AE leading to discontinuation | 48 hours
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-T)] | 48 hours
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] | 48 hours

SECONDARY OUTCOMES:
Number of clinically significant changes in clinical laboratory values, vital signs, ECGs, and physical examinations | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jorn Drappa, Medical Director, Study Director — Alumis Inc
Locations (4):
- United States (4):
  - Advanced Pharma CR, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Undecided
The Sponsor Alumis Inc. is a clinical-stage pharmaceutical company that has not yet adopted an Individual Participant Data (IPD) sharing plan.